CLINICAL TRIAL: NCT05344274
Title: Direct Measures of Retinal Blood Flow and Autoregulation as Robust Biomarkers for Early Glaucoma
Brief Title: Retinal Blood Flow and Autoregulation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Osamah Saeedi, Associate Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-00055126
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma
Keywords: glaucoma; retinal blood flow; erythrocyte mediated angiography; adaptive optics
MeSH Terms: conditions — Glaucoma | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Isocapnic Oxygen (Experimental): Investigators will evaluate retinal blood flow in response to oxygen supplementation.
  Interventions: Diagnostic Test: Indocyanine Green Angiography; Biological: Isocapnic Oxygen; Diagnostic Test: Ocular Imaging with Optical Coherence Tomography (OCT) and Adaptive Optics (AO)

INTERVENTIONS:
Diagnostic Test: Indocyanine Green Angiography — Erythrocyte Mediated Angiography with indocyanine green as well as conventional indocyanine green angiography will be conducted to determine retinal blood flow
Biological: Isocapnic Oxygen — Investigators will evaluate retinal blood flow (RBF) in response to oxygen supplementation at a constant level of carbon dioxide (isocapnic hyperoxia) to isolate the vascular autoregulatory response to oxygen.
Diagnostic Test: Ocular Imaging with Optical Coherence Tomography (OCT) and Adaptive Optics (AO) — Investigators will image subjects with OCT as well as AO technology to determine retinal ganglion cell density, vessel density, and vessel flowrates

SUMMARY:
The purpose of this study is to establish autoregulation of retinal blood flow in arterioles and capillaries as a biomarker for early primary open angle glaucoma.

DETAILED DESCRIPTION:
There is strong evidence for a vascular component in the development and progression of primary open angle glaucoma (POAG). Specifically, glaucoma is associated with impaired retinal blood flow (RBF) and autoregulation of RBF. Autoregulatory impairment may precede retinal ganglion cell (RGC) loss and has been proposed as a potentially early, reversible biomarker. The rationale underlying this proposal is that highly precise and accurate, direct measures of RBF are necessary to study dynamic changes in RBF and their effect on RGCs. Current methods of quantifying RBF remain limited as the majority of imaging modalities provide indirect, relative measurements of RBF. The investigators will directly measure RBF using two robust direct measures: erythrocyte mediated angiography flowmetry (EMAf) and multimodal adaptive optics (mAO). Both techniques allow for the highly accurate and precise measurement of RBF down to the capillary level in the human eye in vivo. The investigators hypothesize that these direct measures of determining absolute RBF will show impaired autoregulation of microvascular RBF in early glaucoma and that this will correlate with glaucomatous damage. The research program will test this hypothesis through two specific aims. In Specific Aim 1, the investigators will determine the extent of impaired autoregulation associated with early glaucoma and measure its ability to predict further glaucoma damage. In Specific Aim 2, the investigators will determine the relationship of capillary density and RGC density in glaucoma subjects and controls. The investigators predict that early glaucoma subjects will exhibit significant measurable impaired vascular autoregulation as compared to controls and that local changes in these parameters will predict structural glaucomatous deficits.

ELIGIBILITY:
Inclusion Criteria:

1. age over 18 years
2. open angle in gonioscopy (grade 3 or 4 in Shaffer classification)
3. refractive error within the range of +3.00 to -8.00 diopters (4) best-corrected visual acuity 20/25 or better (5) Individuals recruited will be in one of the 3 groups:

1) Early Glaucoma as per Hodapp-Anderson-Parrish Criteria (54). Early glaucoma subjects specifically with visual field defects restricted to one side of the horizontal midline will be selected to allow for comparison of rates of progression in both hemifields. Individuals will need to be off of glaucoma medications for four weeks to participate in the study. 2) Pre-perimetric glaucoma defined as the presence of glaucomatous optic nerve damage (e.g., focal notching, rim thinning), RNFL defect, and the absence of a definite glaucomatous visual field defect using standard automated perimetry at the three most recent consecutive examinations. A glaucomatous visual field defect is defined as either 3 or more abnormal points with a P<0.05, of which at least 1 point has a pattern standard deviation (PSD) of P<0.01; or a PSD of P<0.05; or glaucoma hemifield test values outside the normal limits. (55,56) 3) Control group - A subject with no family history of glaucoma who has the following: a) OCT with all four quadrants within the normal range for age-matched controls, b) reliable visual fields with glaucoma hemifield test within normal limits and determined to be normal by a glaucoma specialist, and c) cup-to-disc ratio of 0.4 or lower and asymmetry of the cup to disc ratio no greater than 0.1 as determined by a glaucoma specialist.

Control subjects will be age matched to the early glaucoma subjects.

Exclusion Criteria:

1. corneal abnormalities or other conditions preventing reliable applanation tonometry
2. retinal disease affecting retinal nerve fiber layer thickness such as vitreomacular traction as determined by a glaucoma specialist
3. secondary glaucoma
4. history of prior ocular surgery other than uncomplicated cataract surgery or laser trabeculoplasty
5. inability to safely be off of glaucoma medications for 4 weeks
6. inability to obtain OCT angiography data due to excessive eye motion or inability to fixate
7. unreliable visual fields
8. any history of smoking in the past 6 months
9. cataract greater than lens opacity classification system (LOCS) II Grade≥2
10. diagnosis of diabetes, hypertension, or other known vascular disorder such as vasculitis

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Autoregulation of retinal blood flow | 3 years
  Autoregulation of flow is measured by the percent flow difference in flow between air and oxygen

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland Faculty Physicians, Inc, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Food and Drug Administration (FDA), Silver Spring, Maryland